CLINICAL TRIAL: NCT01284361
Title: User Preference Study to Compare a 40cm Intermittent Catheter to a 30cm Intermittent Catheter
Brief Title: Comparison of Two Intermittent Urinary Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 4875-I
Record Dates: First submitted 2011-01-21; First posted 2011-01-27 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Urinary Retention
Keywords: intermittent catheter; preference
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30 cm Intermittent Catheter (Experimental): Intervention was the test of a 30 cm catheter compared to standard commercial 40 cm catheter in a cross-over design.
  Interventions: Device: 30 cm Intermittent Catheter
- 40 cm Intermittent Catheter (Active Comparator): Active comparator 40 cm commercial catheter was compared to experimental 30 cm catheter in a cross-over design.
  Interventions: Device: 40 cm Intermittent Catheter

INTERVENTIONS:
Device: 30 cm Intermittent Catheter — Randomized cross-over
  Other Names: Apogee Intermittent Catheter
  Arms: 30 cm Intermittent Catheter
Device: 40 cm Intermittent Catheter — randomized cross-over
  Other Names: Apogee Intermittent Catheter
  Arms: 40 cm Intermittent Catheter

SUMMARY:
This is an unblinded, multi-center, randomized, controlled, cross-over study assessing wheel-chair bound, male user preference and catheter characteristics of two intermittent urinary catheters. Subjects enrolled in the study will be randomized to order of catheter use. Individual participation will consist of approximately 1 week of product use. The null hypothesis to be tested is there no difference between catheters.

DETAILED DESCRIPTION:
1. is male and at least 18 years of age.
2. is self-catheterizing at least 3 times a day.
3. has been performing catheterizations for at least 2 months.
4. is wheelchair bound.
5. is able to use a size 12 or 14 French straight catheter.
6. is willing and able to follow the study protocol and Investigator's instructions.
7. is in the opinion of the Investigator, qualified to participate.

ELIGIBILITY:
Inclusion Criteria:

* is male and at least 18 years of age
* is self-catheterizing at least 3 times a day
* has been performing catheterizations for at least 2 months
* wheelchair bound
* is able to use a size 12 or 14 French straight catheter
* is willing and able to follow the study protocol and Investigator's instructions
* is, in the opinion of the Investigator, qualified to participate

Exclusion Criteria:

* has cognitive impairments that preclude completion of study protocol
* cannot communicate as determined by the Investigator
* has an existing medical condition that, in the opinion of the investigator, would interfere with the subject's ability to participate or in the interpretation of the results
* has a symptomatic urinary tract infection determined by interview
* has a retracted penis
* has participated in a study during the previous 30 days involving catheterization
* has been diagnosed with an enlarged prostate
* has urethral strictures, false passages, or urethral obstruction

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Kaurs, MSHSA MT NMT, Study Director — Hollister Incorporated
Locations (4):
- United States (4):
  - Shepherd Center and Crawford Research Institute, Atlanta, Georgia
  - Mark Drug Medical Supply, Wheeling, Illinois
  - Restored Images, Kansas City, Missouri
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Published in Spinal Cord (2013) 51, 772-775

REFERENCES:
- [Result] Costa JA, Menier M, Doran TJ, Kohler TS. Catheter length preference in wheelchair-using men who perform routine clean intermittent catheterization. Spinal Cord. 2013 Oct;51(10):772-5. doi: 10.1038/sc.2013.76. Epub 2013 Jul 30. PMID 23896665
- [Derived] Prieto JA, Murphy CL, Stewart F, Fader M. Intermittent catheter techniques, strategies and designs for managing long-term bladder conditions. Cochrane Database Syst Rev. 2021 Oct 26;10(10):CD006008. doi: 10.1002/14651858.CD006008.pub5. PMID 34699062
- See also: Catheter length preference in wheelchair-using men who perform routine clean intermittent catheterization — http://www.nature.com/sc/journal/v51/n10/full/sc201376a.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: October 10, 2010 - July 21 , 2011 types of locations: private vendor, public rehabilitation center, university
Groups:
- Control and Test Crossover: test and control intermittent urinary catheters : randomized cross-over
Period: Overall Study
Arm/Group | Control and Test Crossover
Started | 91
Completed | 82
Not Completed | 9
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 5
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Each subject was given 10 Control catheters and 10 Test catheters to be used consecutively until all 20 catheters were used. Subjects used either the Test catheters (A) first and then the Control catheters (B) or vice versa. Subjects completed questionnaire after using each catheter and a preference questionnaire after all catheters were used.
Arm/Group | Control and Test Crossover
Number analyzed (Participants) | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 82
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (11.7)
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 82
Region of Enrollment [Number; unit: participants]
  United States | 82

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants
Description: Percentage of participants that preferred the 40 cm catheter
Time Frame: 1 week
Measure: Number; unit: percentage of participants
Groups:
- Control and Test Crossover: Control and test intermittent urinary catheters : randomized cross-over
Arm/Group | Control and Test Crossover
Number analyzed (Participants) | 82
percentage of participants | 91.5
Statistical Analysis 1: Comparison: Control and Test Crossover; The sample size of 81 subjects provides a 10.8% margin of error; Test type: Superiority or Other; Proportion = 91.5, 95% CI 2-sided [84.5 to 97.5] — Seventy five of the 82 subjects (91.5%) preferred the longer commercially available catheter over the experimental 30 cm catheter

2. Secondary Outcome: Assessment of Ease of Use Characteristics
Description: Ease of insertion, removal, and control while catheterizing were assessed using a 5 point Likert scale. The numbers recorded are the percentage of the "top" two responses on a 5 point Likert scale. On one scale this includes 1) Very Easy or 2) Easy, on a scale ranging from 1) Very Easy to 5) Very Difficult. On the other scale this includes 1) Strongly Agree or 2) Agree on a scale ranging from 1) Strongly Agree to 5) Strongly Disagree.
Time Frame: 1 week
Population: 82 self-catheterizing wheelchair-using men
Measure: Number; unit: percentage of participants
Groups:
- Control 40 cm Catheter: Commercial gel lubricated 40 cm catheter
- Test 30 cm Catheter: Test gel lubricated 30 cm catheter identical in all aspects to Control catheter except being 10 cm shorter
Arm/Group | Control 40 cm Catheter | Test 30 cm Catheter
Number analyzed (Participants) | 82 | 82
percentage of participants
  Ease of insertion | 84.65 | 67.78
  Ease of Removal | 94.85 | 86.34
  Ease of Catheter Control Upon Urethral Insertion | 86.48 | 72.19
  Confidence of Complete Bladder Drainage | 84.15 | 45.80
  Ease of Draining into Receptacle | 87.00 | 58.02
  Ease of Connecting Urine Bag | 35.68 | 31.49

ADVERSE EVENTS:
Groups:
- Control 40 cm Catheter: Commercial 40 cm gel lubricated catheter
- Test 30 cm Catheter: Test 30 cm gel lubricated cather similar in all aspects except 10 cm shorter length as control catheter
Arm/Group | Control 40 cm Catheter | Test 30 cm Catheter
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/91
Other Adverse Events (participants affected / at risk) | 0/91 | 2/91
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control 40 cm Catheter (N=91) | Test 30 cm Catheter (N=91)
bleeding (Renal and urinary disorders) | 0 (0) | 1 (91) — reported mild urethral bleeding after using one 30 cm catheter
discomfort (Renal and urinary disorders) | 0 (0) | 1 (91) — reported mild pain when he used all ten 30 cm catheters

LIMITATIONS AND CAVEATS:
Male catheter users only in USA only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Variable restriction depends on site.